CLINICAL TRIAL: NCT06106334
Title: A Crossover, Phase 1, Open-label, One-arm Study to Investigate the Effect of Itraconazole on the Pharmacokinetics of S-309309 in Healthy Male and Female Participants
Brief Title: Effect of Administration of Itraconazole on the Pharmacokinetics of S-309309 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2301N1113
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Healthy Volunteers
MeSH Terms: conditions — Obesity | interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- S-309309 (Experimental): All participants will receive each of the following treatments:
  * Days 1 and 19: S-309309 once daily (QD); in the fasted state)
  * Day 15: Itraconazole twice daily (BID); in the fed state)
  * Days 16 to 24: Itraconazole QD (in the fed state, except for Day 19 [co-administration with S-309309 in the fasted state])
  Interventions: Drug: S309309; Drug: Itraconazole

INTERVENTIONS:
Drug: S309309 — Administered as oral capsules
Drug: Itraconazole — Administered as oral capsules

SUMMARY:
The primary purpose of this study is to determine the effect of repeated administration of itraconazole on the pharmacokinetic (PK) profile of S-309309; and the PK of S-309309 following administration of S-309309 alone and co-administration with itraconazole

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who are considered to be medically healthy as determined by the investigator
* Participants whose body mass index (BMI) is within the range of ≥ 18.5 to ≤ 30.0 kg/m^2
* Contraceptive use by male and female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Participants who understand the study procedures and agree to participate by providing written informed consent
* Participants who are willing and able to comply with all study procedures and restrictions

Key Exclusion Criteria:

* Participants who have a history of clinically significant hypersensitivity or severe side effects induced by a drug.
* Participants who have a history of ventricular dysfunction, congestive heart failure, or pulmonary edema.
* Participants who have a history of gastrointestinal surgery including, but not limited to, cholecystectomy, gastric resection, and/or intestinal resection that may result in a clinically significant abnormality in gastrointestinal function (except for an appendectomy). Participants can be considered by the investigator (or sub-investigator) to be ineligible for the study due to a history of or current condition of significant metabolic or endocrine, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, immunological, neurological, or psychiatric disorders with clinical manifestations.
* Participants who are considered inappropriate for participation in the study for any reason by the investigator (or sub-investigator).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve Extrapolated From Time 0 to Infinity (AUC0-inf) After Administration of S-309309 | Up to 2 weeks postdose on Days 1, 19
Area Under the Concentration-Time Curve Extrapolated From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) After Administration of S-309309 | Up to 2 weeks postdose on Days 1, 19
Maximum Observed Plasma Concentration (Cmax) After Administration of S-309309 | Up to 2 weeks postdose on Days 1, 19

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Shionogi
Locations (1):
- Fortrea Clinical Research Unit Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No